CLINICAL TRIAL: NCT04963660
Title: CASE SERIES OF PRIMARY IMMUNODEFICIENCIES IN ADULTS DIAGNOSED IN TWO HOSPITALS OF THE TERTIARY LEVEL OF CARE OF THE COSTA RICAN SOCIAL SECURITY Fund, 2017-2018
Brief Title: Primary Immunodeficiencies in Costa Rican Adults
Status: Completed | Type: Observational
Sponsor: Caja Costarricense de Seguro Social (Other Government)
Responsible Party: Sponsor
Other Study IDs: R017-SABI-00148.
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Primary Immune Deficiency in Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary immunodeficiencies represent a underdiagnosed group of rare diseases which if diagnosed well and in time can be treated in an efficient manner and prevent complications that may affect the quality of patients life in an severe manner. Neither in Costa Rica nor in Central America studies or national registries regarding the prevalence and characterization of primary immunodeficiencies in adult patients exist up to now. This study reflects for the first time the epidemiologic situation of primary immunodeficiencies in a Central American country, characterizing adult patients diagnosed with primary and idiopathic immune disorders treated in two specialized immunodeficiency clinics in Costa Rica.

ELIGIBILITY:
Inclusion Criteria:

* All patients from adult primary immunodeficiency clinics will be included.

Exclusion Criteria:

* Patients with HIV
* Proven secondary immunodeficiencies.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cases of primary immunodeficiency and idiopathic defects of immunity detected in the primary immunodeficiency clinics of the Hospitals Mexico and Dr. Rafael Ángel Calderón Guardia between November 2017 and May 2018.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Clinical manifestations of all adult patients diagnosed with primary and idiopathic immune defects | 1 year
  Describe the clinical manifestations of all adult patients diagnosed with primary and idiopathic immune defects attended in the primary immunodeficiency clinics of the Hospitals Mexico and Dr. Rafael Ángel Calderón Guardia during the study period.

SECONDARY OUTCOMES:
characterization of immunodeficient patients | 1 year
  Characterize immunodeficient patients using sociodemographic and health variables.
Concordances between clinical manifestations and literature | 1 year
  •Establish concordances between the clinical manifestations of the group of patients under study with those described in the literature according to the different pathologies.
organic complications | 1 year
  Record organic complications secondary to immunodeficiency status.
type and degree of immunodeficiency | 1 year
  Differentiate the type and degree of immunodeficiency of each patient.
pathonges that cause infectious | 1 year
  Report isolated pathogens that cause infectious manifestations in patients.
bacteria present in upper airways | 1 year
  •Report the colonizing bacteria present in the cultures of the upper airways of the patients requested in the initial approach.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Calderon Guardia, San José, Costa Rica